CLINICAL TRIAL: NCT05603273
Title: Non-weight Bearing Exercise for Accelerated Healing of Diabetic Foot Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jacob Haus, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00202034; DISP (Other Grant/Funding Number: University of Michigan)
Record Dates: First submitted 2022-10-26; First posted 2022-11-02 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Type2diabetes; Foot Ulcer
MeSH Terms: conditions — Foot Ulcer

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard wound care (No Intervention): normal wound care according to current clinical practice
- non-weight bearing exercise + standard wound care (Experimental): normal wound care according to current clinical practice with the addition of a weekly exercise routine
  Interventions: Behavioral: non-weight bearing exercise

INTERVENTIONS:
Behavioral: non-weight bearing exercise — exercise on a non-weight bearing device at 50% of peak capacity, 3 days per week for 6 weeks
  Arms: non-weight bearing exercise + standard wound care

SUMMARY:
The goal of this study is to improve the therapeutic management of diabetic foot ulcers (DFU). The main questions to answer are if a program of non-weight bearing exercise helps the DFU heal faster than standard wound care. This randomized clinical trial will determine how blood flow to the ulcer and whole body metabolism may be improved with exercise. Participants will be randomized to either exercise + standard wound care or standard wound care alone and undergo testing for leg blood flow, fitness and measures of metabolism through blood draws. The intervention period is 6-weeks. Eligible participants must have an existing foot ulcer uncomplicated by infection and be medically cleared to exercise.

DETAILED DESCRIPTION:
This research is being done because people with diabetes have reduced healing capacity. This can be problematic because wounds that do not heal may turn into ulcers which may lead to more severe complications. Non-weight bearing exercise has many positive health benefits that improve metabolic and vascular health which will then improve healing time. Therefore, the purpose of this study is to evaluate the positive effects of non-weight bearing exercise. Once the effects of non-weight bearing exercise are confirmed, progress towards the prevention and treatment of diabetic foot ulcers and complications may be possible. Potential participants are eligible for the study if diagnosed with type 2 diabetes and have a foot ulcer or wound. Approximately 40 subjects with Type 2 Diabetes are expected to complete this study. Participation in this study requires medical clearance following a screening visit and then being randomly assigned to a non-weight bearing exercise training group or a control group. Both groups will receive standard diabetic and wound care. Subjects will complete 7 study visits at the University of Michigan. The research tests during these visits will include measures of body composition, oral glucose tolerance test, exercise testing, blood draws, vascular function measurements, wound measurement, single-leg exercise session and group randomization If randomized to the Exercise Group subjects will be asked to visit the University of Michigan three days a week for 6 weeks. During each visit during this 6-week period, subjects will perform exercise training by completing 30 minutes of single-leg exercise at approximately 50% of a predetermined maximal effort. Regardless of the group subjects are randomized to, all will receive standard care for the management of diabetes foot ulcer/wound.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or Female, aged 18 yrs or older
4. Diabetes diagnosed or meets ADA criteria for Type 2 diabetes
5. Foot ulcer of diabetic etiology, with all of the following characteristics:

   * Ulcer size > 0.5cm2 and < 12cm2 at least 2 cm from any other ulcer
   * Ulcer with Wagner grade 1 or 2
6. In case of multiple ulcers, select the largest ulcer that meets inclusion criteria.

Exclusion Criteria:

1. Patient participating in an interventional clinical trial within 1 month of visit 1
2. Participant has Charcot's foot or other foot deformities that prevent adequate targeted ulcer offloading
3. Participant has active severe infection or osteomyelitis at the time of the screening visit
4. History of cancer within the last 3 years, other than non-melanoma skin cancer
5. Use of adjunctive therapy within previous 30 days
6. Currently receiving medication considered to be a systemic glucocorticoid
7. Plan to perform a vascular intervention, such as surgical bypass, angioplasty or stenting, or < 1 month from a prior ipsilateral (same side) vascular intervention
8. Pregnant or currently lactating
9. Uncontrolled blood glucose with presence of urinary ketones
10. Contraindications for exercise as define by the American Heart Association/American College of Sports Medicine Guidelines for Exercise Testing and Prescription [1]
11. Bilateral wound or ulcer
12. Current infection of COVID19
13. Any history of concomitant medical condition that, in the opinion of the investigator(s), would compromise the participants ability to safely complete the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
wound size and depth | 6 weeks
  wound site and depth

SECONDARY OUTCOMES:
blood flow | 6 weeks
  blood flow by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Haus, PhD, Principal Investigator — University of Michigan
Locations (1):
- School of Kinesiology, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
no plan to share data at this time